CLINICAL TRIAL: NCT00491478
Title: Stereotypies and Mental Retardation: Neurobiological Basis
Brief Title: Repetitive Behavior Disorders in People With Severe Mental Retardation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: R01HD030615 (NIH)
Record Dates: First submitted 2007-06-22; First posted 2007-06-26 (Estimated); Last update posted 2007-06-26 (Estimated); Status verified 2003-05

CONDITIONS: Mental Retardation; Stereotyped Behavior; Self-Injurious Behavior; Compulsive Behavior
Keywords: Repetitive behavior disorder; Stereotypy; Sertraline
MeSH Terms: conditions — Intellectual Disability; Stereotyped Behavior; Self-Injurious Behavior; Compulsive Behavior; Stereotypic Movement Disorder | interventions — Sertraline

INTERVENTIONS:
Drug: sertraline

SUMMARY:
Repetitive behavior disorders are prevalent among people with severe mental retardation. These disorders can interfere significantly with an individual's daily functions. This trial is part of a long-term project that has studied the biologic basis of and possible treatments for repetitive behavior disorders. The trial will evaluate the effectiveness of two medications, a selective serotonin reuptake inhibitor (SSRI) and an atypical antipsychotic, in treating repetitive behavior disorders in people with mental retardation.

DETAILED DESCRIPTION:
Abnormal repetitive behaviors (odd or inappropriate movements, self-injury, and compulsions) are among the aberrant behaviors exhibited by individuals with mental retardation. However, little is known about their pathobiology and treatments are largely unconfirmed by controlled trials. For example, few controlled studies have examined the efficacy of pharmacological treatment of abnormal repetitive behavior in individuals with mental retardation.

This trial is part of a larger project designed to elucidate the neurobiological bases of repetitive behavior disorders and to develop rational, safe, and effective pharmacological treatments. Thus far, the project has established a pathophysiological basis for stereotyped behavior disorder, demonstrated the role of central dopamine deficiency in stereotyped behavior disorder, and provided evidence of the efficacy of both 5-HT uptake inhibitors and atypical antipsychotics in treating stereotyped behaviors.

There is currently little information to guide the clinician in deciding which drug class may be more effective for which abnormal repetitive behaviors and for which individuals. Moreover, little work has attempted to identify variables that may predict differential treatment response. This trial will assess the relative efficacy of an SSRI and an atypical antipsychotic across multiple categories of abnormal repetitive behaviors.

ELIGIBILITY:
Inclusion Criteria

* Mental retardation
* Medically stable resident of either Western Carolina Center, Morganton, NC or Tacachale Community, Gainesville, FL
* Free of sensory deficits
* Ambulatory
* High rate of stereotyped behavior that may co-occur with self-injurious or compulsive behaviors

Exclusion Criteria

* Poor general health
* Cardiac, hepatic, or renal abnormalities
* Seizure within 4 months prior to study entry (patients on seizure medication who have not had a seizure within 4 months prior to study entry may participate)
* Tardive dyskinesia
* Akathisia
* Neuroleptic use within 6 months of study entry
* History of sensitivity to ergot alkaloids
* Hypertension

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1992-09

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lewis, PhD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - Department of Psychiatry, Gainesville, Florida
  - Western Carolina Center, Morganton, North Carolina

REFERENCES:
- [Background] Bodfish JW, Crawford TW, Powell SB, Parker DE, Golden RN, Lewis MH. Compulsions in adults with mental retardation: prevalence, phenomenology, and comorbidity with stereotypy and self-injury. Am J Ment Retard. 1995 Sep;100(2):183-92. PMID 8527113
- [Background] Lewis MH, Bodfish JW, Powell SB, Wiest K, Darling M, Golden RN. Plasma HVA in adults with mental retardation and stereotyped behavior: biochemical evidence for a dopamine deficiency model. Am J Ment Retard. 1996 Jan;100(4):413-8. No abstract available. PMID 8718995
- [Background] Bodfish JW, Symons FJ, Parker DE, Lewis MH. Varieties of repetitive behavior in autism: comparisons to mental retardation. J Autism Dev Disord. 2000 Jun;30(3):237-43. doi: 10.1023/a:1005596502855. PMID 11055459
- [Background] Bodfish JW, Parker DE, Lewis MH, Sprague RL, Newell KM. Stereotypy and motor control: differences in the postural stability dynamics of persons with stereotyped and dyskinetic movement disorders. Am J Ment Retard. 2001 Mar;106(2):123-34. doi: 10.1352/0895-8017(2001)1062.0.CO;2. PMID 11321603